CLINICAL TRIAL: NCT01643993
Title: Intrauterine Human Chorionic Gonadotropin at the Time of Embryo Transfer: A Randomized Controlled Trial
Brief Title: Intrauterine Human Chorionic Gonadotropin at the Time of Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMA-2012-01
Record Dates: First submitted 2012-06-28; First posted 2012-07-18 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Control Media Only; Study hCG and Media
Keywords: IVF; embryo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hCG at Time of Embryo Transfer (Experimental): Patients will have hCG and media (for a total of 20 microliters) inserted during a mock embryo transfer immediately prior to actual embryo transfer.
  Interventions: Other: hCG at the Time of Embryo Transfer
- Control (Other): Patients will have 20 microliters of media inserted during a mock embryo transfer immediately prior to actual embryo transfer.
  Interventions: Other: Control

INTERVENTIONS:
Other: hCG at the Time of Embryo Transfer — hCG will be included in the 20 microliters of media inserted during a mock embryo transfer immediately prior to actual embryo transfer.
  Arms: hCG at Time of Embryo Transfer
Other: Control — Patients will have 20 microliters of media inserted during a mock embryo transfer immediately prior to actual embryo transfer.
  Arms: Control

SUMMARY:
Techniques to improve pregnancy and delivery rates in IVF cycles have focused not only on the embryos transferred, but also the conditions in the uterus at the time of transfer and implantation. Prior studies have shown that embryos secrete human chorionic gonadotropin (hCG) prior to implantation. However, in IVF cycles, the embryos have limited time to secrete hCG before implantation must occur because embryos are placed into the uterus rather than traveling there from the fallopian tubes. Recent studies have shown that the introduction of hCG into the uterus prior to embryo transfer may make the uterus more receptive to implantation. These studies involved day 3 embryos and the investigators are seeking to evaluate the potential benefits of hCG on implantation rates of blastocysts (day 5 or day 6 embryos).

The purpose of this study is to determine whether infusion of human chorionic gonadotropin (hCG) into the uterus immediately prior to embryo transfer results in increased implantation rates.

The entire IVF cycle, fresh or frozen, will be conducted per routine. All laboratory culture conditions will be per routine. In fresh and frozen IVF cycles, an embryo transfer will be performed per routine.

At the time of embryo transfer, participants will be randomly assigned to either the control group or the hCG group. Patients in the hCG group will have a mock embryo transfer with 20µL of transfer media including 500IU of hCG. Patients in the control group will have a mock embryo transfer with 20µL of transfer media.

All post-transfer care and pregnancy monitoring will be identical and per routine protocol.

ELIGIBILITY:
Inclusion Criteria:

* all patients 43 years old or under undergoing fresh or frozen IVF cycles are eligible to participate

Exclusion Criteria:

* patients greater than 43 years old
* patinets currently participating in any other research studies

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Sustained implantation rate | 12 weeks
  Sustained implantation rate is measured as the number of fetal heart beats seen at the time of patient discharge to OB/GYN care (approximately 8 weeks gestation).

SECONDARY OUTCOMES:
Ongoing pregnancy rate | 9 Weeks
  The number of pregnancies with at least one fetal heart beat seen at the time of discharge to OB/GYN care per embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (2):
- United States (2):
  - Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey
  - Reproductive Medicine Associates of Pennsylvania at Lehigh Valley, Allentown, Pennsylvania

REFERENCES:
- [Derived] Hong KH, Forman EJ, Werner MD, Upham KM, Gumeny CL, Winslow AD, Kim TJ, Scott RT Jr. Endometrial infusion of human chorionic gonadotropin at the time of blastocyst embryo transfer does not impact clinical outcomes: a randomized, double-blind, placebo-controlled trial. Fertil Steril. 2014 Dec;102(6):1591-5.e2. doi: 10.1016/j.fertnstert.2014.08.006. Epub 2014 Sep 16. PMID 25234040